CLINICAL TRIAL: NCT04105023
Title: Genistein Stimulates Insulin Sensitivity Through Gut Microbiota Reshaping and Skeletal Muscle AMPK Activation in Obese Subjects
Brief Title: Genistein Stimulates Insulin Sensitivity Through Gut Microbiota
Acronym: GENISTEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Armando Tovar, Lab Director and Senior Scientist of the department of nutrition physiology, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1099
Record Dates: First submitted 2019-09-20; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: genistein; gut microbiota; AMPK; fatty acid oxidation
MeSH Terms: conditions — Metabolic Syndrome; Obesity | interventions — Genistein

STUDY DESIGN:
Intervention Model Description: These individuals were advised to consume the recommended diet for subjects with MetS according to the guidelines of the ATPIII. Patients were randomly distributed to consume a) placebo treatment or b) genistein capsules (50 mg/day). The participants were followed for 2 months
Who Masked: Participant, Investigator
Masking Description: The interventions with genistein and placebo were identically encapsulated in appearance, both the researcher and the participant did not know what type of maneuver was assigned. The bottle with the capsules was distributed by a person outside the study who was the same one who performed the randomization.
  Study staff and participants were blinded during the assignment and execution of the interventions in the study. the capsules delivered to the participants were 2 per day, the capsules had the same color and appearance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- genistein (Experimental): Genistein capsules of 25 mg each, 50mg/day
  Interventions: Dietary Supplement: genistein
- placebo (Placebo Comparator): Maltodextrin capsules, administered orally once every 12 hours
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: genistein — Administered orally once every 12 hours
  Arms: genistein
Dietary Supplement: Placebo — Administered orally once every 12 hours
  Arms: placebo

SUMMARY:
There is evidence that genistein present in soy can improve insulin resistance in rodents and humans with metabolic syndrome (MetS). However, it is not known if this improvement is associated with changes in the gut microbiota. In the present study, the investigators show that the consumption of genistein for 2 months could have an effect on insulin resistance in subjects with MetS. This effect will be accompanied by a modification of the gut microbiota taxonomy. As a consequence, there will be a reduction in metabolic endotoxemia accompanied by an increase in AMP-activated protein kinase (AMPK) phosphorylation and the expression of genes of fatty acid oxidation in skeletal muscle.

DETAILED DESCRIPTION:
The investigators included 45 participants who met the following inclusion criteria: adults between 20 and 60 years of age with a diagnosis of MetS, HOMA index greater than 2.5, BMI ≥30 and ≤ 40 kg / m2 and who signed the consent letter. Patients who had any added pathology, pregnancy, smoking or consumed medications were excluded. Once the letter of informed consent was accepted, the patients were assigned to the respective treatment group. These individuals were advised to consume the recommended diet for subjects with MetS according to the guidelines of the ATPIII. Participants were randomly distributed to consume a) placebo treatment or b) genistein capsules (50 mg/day). The participants were followed for 2 months. In the previsit, informed consent letters were given, and blood samples were taken to evaluate glucose concentration, lipid profile, lipopolysaccharide and serum insulin. Also determined blood pressure, body weight, height, body composition and gut microbiota. The presence of insulin resistance was determined by means of the HOMA-IR index and by an oral glucose tolerance test. After 2 months, the same variables were assessed, and an expert surgeon in the operating room performed a vastus lateralis muscle biopsy, then RNA extraction and gene expression microarray assay was performed

ELIGIBILITY:
Inclusion Criteria:

* Adults (men and women) between the ages of 18 and 50.
* Patients with obesity (BMI ≥ 30 and ≤ 40 kg / m2) and with insulin resistance (HOMA - IR Index ≥ 2.5).
* Mexican mestizos (parents and grandparents born in Mexico).
* Patients who can read and write.

Exclusion Criteria:

* • Patients with any type of diabetes.

  * Patients with kidney disease diagnosed by a medical or with creatinine> 1.3 mg / dL for men and > 1.1 mg / dL for women and / or BUN> 20 mg / dL.
  * Patients with acquired diseases that produce obesity and diabetes secondarily.
  * Patients who have suffered a cardiovascular event.
  * Patients with weight loss > 3 kg in the last 3 months.
  * Patients with any catabolic diseases.
  * Gravidity status
  * Positive smoking
  * Treatment with any medication

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-09-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
intestinal microbiota | Baseline to 2 month
  Measurement of gut microbiota by sequencing using the Illumina platform

SECONDARY OUTCOMES:
glucose metabolism profile | Baseline to 2 month
  serum glucose (mg/dL)
Glucose metabolism profile | Baseline to 2 month
  serum insulin (µUI/ml)
Triglycerides | Baseline to 2 month
  serum triglycerides (mg/dL)
Total Cholesterol | Baseline to 2 month
  serum total cholesterol (mg/dL)
LDL cholesterol | Baseline to 2 month
  serum LDL cholesterol (mg/dL)
HDL cholesterol | Baseline to 2 month
  serum HDL cholesterol (mg/dL)
Inflammatory profile | Baseline to 2 month
  plasma lipopolysaccharide (LPS) (ng/mL)
Body weight | Baseline to 2 month
  body weight (kg)
Blood pressure | Baseline to 2 month
  blood pressure (mmHg)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guevara-Cruz M, Flores-Lopez AG, Aguilar-Lopez M, Sanchez-Tapia M, Medina-Vera I, Diaz D, Tovar AR, Torres N. Improvement of Lipoprotein Profile and Metabolic Endotoxemia by a Lifestyle Intervention That Modifies the Gut Microbiota in Subjects With Metabolic Syndrome. J Am Heart Assoc. 2019 Sep 3;8(17):e012401. doi: 10.1161/JAHA.119.012401. Epub 2019 Aug 27. PMID 31451009
- [Background] Palacios-Gonzalez B, Vargas-Castillo A, Velazquez-Villegas LA, Vasquez-Reyes S, Lopez P, Noriega LG, Aleman G, Tovar-Palacio C, Torre-Villalvazo I, Yang LJ, Zarain-Herzberg A, Torres N, Tovar AR. Genistein increases the thermogenic program of subcutaneous WAT and increases energy expenditure in mice. J Nutr Biochem. 2019 Jun;68:59-68. doi: 10.1016/j.jnutbio.2019.03.012. Epub 2019 Mar 29. PMID 31030168
- [Background] Lopez P, Sanchez M, Perez-Cruz C, Velazquez-Villegas LA, Syeda T, Aguilar-Lopez M, Rocha-Viggiano AK, Del Carmen Silva-Lucero M, Torre-Villalvazo I, Noriega LG, Torres N, Tovar AR. Long-Term Genistein Consumption Modifies Gut Microbiota, Improving Glucose Metabolism, Metabolic Endotoxemia, and Cognitive Function in Mice Fed a High-Fat Diet. Mol Nutr Food Res. 2018 Aug;62(16):e1800313. doi: 10.1002/mnfr.201800313. Epub 2018 Jul 29. PMID 29979819
- [Background] Medina-Vera I, Sanchez-Tapia M, Noriega-Lopez L, Granados-Portillo O, Guevara-Cruz M, Flores-Lopez A, Avila-Nava A, Fernandez ML, Tovar AR, Torres N. A dietary intervention with functional foods reduces metabolic endotoxaemia and attenuates biochemical abnormalities by modifying faecal microbiota in people with type 2 diabetes. Diabetes Metab. 2019 Apr;45(2):122-131. doi: 10.1016/j.diabet.2018.09.004. Epub 2018 Sep 25. PMID 30266575